CLINICAL TRIAL: NCT01007721
Title: Randomised, Double-blind, Triple Dummy, Partial Cross-over (Each Active Treatment With Placebo) Study Using an Environmental Challenge Chamber (ECC) to Assess the Safety and Efficacy of 2 Weeks of Oral BI 671800 ED 50, 200 or 400 mg Bid, Compared to Montelukast 10 mg qd, Fluticasone Propionate Nasal Spray 200 µg qd (2 Nasal Actuations Each Nostril of 50 µg) Versus Placebo in Seasonal Allergic Rhinitis Patients Out of Season, Sensitive to Dactylis Glomerata.
Brief Title: Randomized, Placebo Controlled, Crossover Study in an Environmental Challenge Chamber to Assess Safety & Efficacy of Three Oral Doses of BI 671800 Versus Fluticasone Propionate and Montelukast in Sensitive Seasonal Allergic Rhinitis Patients Out of Season
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1268.41; 2009-013269-24
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Rhinitis, Allergic, Seasonal; Asthma
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Asthma | interventions — montelukast; Tablets

ARMS (6):
- BI 671800 ED 100 mg (Experimental): 2 capsules of BI 671800 ED 25 mg plus 2 capsules of BI 671800 ED placebo (bid in the morning and evening) plus 1 over-encapsulated montelukast placebo tablet (qd in the morning) plus fluticasone propionate placebo nasal spray (2 puffs each nostril qd in the morning)
  Interventions: Drug: BI 67100 ED 25 mg; Drug: BI 671800 ED placebo; Drug: montelukast placebo tablet; Drug: fluticasone propionate placebo nasal spray
- BI 671800 ED 400 mg (Experimental): 2 capsules of BI 671800 ED 100 mg plus 2 capsules of placebo (bid in the morning and evening) plus 1 over-encapsulated montelukast placebo tablet (qd in the morning) plus fluticasone propionate nasal spray placebo (2 puffs each nostril qd in the morning)
  Interventions: Drug: fluticasone propionate placebo nasal spray; Drug: BI 671800 ED 100 mg; Drug: 671800 ED placebo; Drug: montelukast placebo tablet
- Montelukast 10 mg (Active Comparator): 1 over-encapsulated montelukast 10 mg tablet (qd in the morning) plus 4 capsules of BI 671800 ED placebo (bid in the morning and evening) plus fluticasone propionate placebo nasal spray (2 puffs each nostril qd in the morning)
  Interventions: Drug: fluticasone propionate placebo nasal spray; Drug: BI 671800 ED placebo; Drug: montelukast 10 mg tablet
- Fluticasonepropionate nasal spray 200¿g (Active Comparator): Fluticasonepropionate nasal spray 200 mcg (qd, 2 puffs of 50 ¿g per nostril) plus 4 capsules of BI 671800 ED placebo (bid in the morning and evening) plus 1 overencapsulated montelukast placebo tablet (qd in the morning)
  Interventions: Drug: BI 671800 ED placebo; Drug: montelukast placebo tablet; Drug: Fluticasonepropionate nasal spray 200 mcg
- BI 671800 ED placebo (Placebo Comparator): 4 capsules of BI 671800 ED placebo (bid in the morning and evening), plus 1 over-encapsulated montelukast placebo tablet (qd in the morning) plus fluticasone propionate placebo nasal spray (2 puffs each nostril qd in the morning)
  Interventions: Drug: montelukast placebo tablet; Drug: BI 671800 ED placebo; Drug: fluticasone propionate placebo nasal spray
- BI 671800 ED 800 mg (Experimental): 4 capsules of BI 671800 ED 100 mg (bid in the morning and evening) plus 1 over-encapsulated montelukast placebo tablet (qd in the morning) plus fluticasone propionate nasal spray placebo (2 puffs each nostril qd in the morning)
  Interventions: Drug: BI 671800 ED 100 mg; Drug: montelukast placebo tablet; Drug: fluticasone propionate nasal spray placebo

INTERVENTIONS:
Drug: BI 67100 ED 25 mg — 2 capsules of BI 671800 ED 25 mg
  Arms: BI 671800 ED 100 mg
Drug: BI 671800 ED placebo — 2 capsules of BI 671800 ED placebo (bid in the morning and evening)
  Arms: BI 671800 ED 100 mg
Drug: montelukast placebo tablet — 1 over-encapsulated montelukast placebo tablet (qd in the morning)
  Arms: BI 671800 ED 100 mg
Drug: montelukast placebo tablet — 1 over-encapsulated montelukast placebo tablet (qd in the morning)
  Arms: BI 671800 ED placebo
Drug: fluticasone propionate placebo nasal spray — fluticasone propionate placebo nasal spray (2 puffs each nostril qd in the morning)
  Arms: BI 671800 ED 100 mg
Drug: fluticasone propionate placebo nasal spray — fluticasone propionate placebo nasal spray (2 puffs each nostril qd in the morning)
  Arms: BI 671800 ED 400 mg
Drug: fluticasone propionate placebo nasal spray — fluticasone propionate placebo nasal spray (2 puffs each nostril qd in the morning)
  Arms: Montelukast 10 mg
Drug: BI 671800 ED 100 mg — 4 capsules of BI 671800 ED 100 mg (bid in the morning and evening)
  Arms: BI 671800 ED 800 mg
Drug: BI 671800 ED placebo — 4 capsules of BI 671800 ED placebo (bid in the morning and evening)
  Arms: Montelukast 10 mg
Drug: BI 671800 ED placebo — 4 capsules of BI 671800 ED placebo (bid in the morning and evening)
  Arms: BI 671800 ED placebo
Drug: BI 671800 ED placebo — 4 capsules of BI 671800 ED placebo (bid in the morning and evening)
  Arms: Fluticasonepropionate nasal spray 200¿g
Drug: BI 671800 ED 100 mg — 2 capsules of BI 671800 ED 100 mg (bid in the morning and evening)
  Arms: BI 671800 ED 400 mg
Drug: 671800 ED placebo — 2 capsules of BI 671800 ED placebo (bid in the morning and evening)
  Arms: BI 671800 ED 400 mg
Drug: montelukast placebo tablet — 1 over-encapsulated montelukast placebo tablet (qd in the morning)
  Arms: BI 671800 ED 400 mg
Drug: montelukast placebo tablet — 1 over-encapsulated montelukast placebo tablet (qd in the morning)
  Arms: BI 671800 ED 800 mg
Drug: montelukast placebo tablet — 1 over-encapsulated montelukast placebo tablet (qd in the morning)
  Arms: Fluticasonepropionate nasal spray 200¿g
Drug: montelukast 10 mg tablet — 1 over-encapsulated montelukast 10 mg tablet (qd in the morning)
  Arms: Montelukast 10 mg
Drug: fluticasone propionate placebo nasal spray — fluticasone propionate placebo nasal spray (2 puffs each nostril qd in the morning)
  Arms: BI 671800 ED placebo
Drug: fluticasone propionate nasal spray placebo — fluticasone propionate nasal spray placebo (2 puffs each nostril qd in the morning)
  Arms: BI 671800 ED 800 mg
Drug: Fluticasonepropionate nasal spray 200 mcg — Fluticasonepropionate nasal spray 200 mcg (qd, 2 puffs of 50 mcg per nostril)
  Arms: Fluticasonepropionate nasal spray 200¿g

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of BI 671800 ED using three dose levels of BI 671800 ED (50 mg, 200 mg and 400 mg), administered twice daily compared to FP (fluticasone propionate) nasal 100 mcg per nostril qd in the morning or Montelukast 10 mg qd am given for 2 weeks in patients with SAR (seasonal allergic rhinitis) out of season using an environmental exposure chamber in patients known to be sensitive to the aero-allergen Dactylis glomerata.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent consistent with ICH-GCP guidelines (International Conference on Harmonisation for Good Clinical Practice) and local legislations prior to any study-related procedures, which includes medication washout and restrictions.
2. Male or female, with a diagnosis of seasonal allergic rhinitis by a physician with a positive skin prick test to Dactylis glomerata within 12 months prior to Visit 2
3. TNSS (total nasal symptom score) of less or equal than 2 before start of challenge at Visit 2 and a TNSS of > 5 at least once during the 2h-baseline ECC exposure
4. 18 to 65 years of age (age inclusive)
5. Non-smoker or ex-smoker with a cigarette smoking history of less or equal than 10 pack-years (and smoking cessation for at least one year prior to enrolment) with negative urinary cotinine at screening (Visit 1)
6. Ability to comply with requirements, medication restrictions (see 4.2.2) and procedures of the study protocol including AM1® device and rescue medication use.
7. Pre-bronchodilator FEV1 (forced expiratory volume in one second) equal or greater than 80% of predicted value (European Community for Steel and Coal) at screening
8. BMI between 18 and 35 (Body Mass Index)
9. Negative breath -alcohol, urine -cotinine and -drug tests at screening (Visit 1)

Exclusion Criteria:

1. Significant pulmonary disease other than allergic rhinitis (or mild intermittent asthma managed by SABA (short acting bronchodilator) alone) or other medical conditions* that may, in the opinion of the investigator result in the any of the following:

   * put the patient at risk because of participation in the study
   * influence the results of the study (as determined by medical history, examination and clinical investigations at screening)
   * cause concern regarding the patient's ability to participate in the study. *e.g. cardiac, gastro-intestinal, hepatic, renal, metabolic, dermatologic, neurological, haematological, oncological and psychiatric. Patients with malignancy for which the patient has undergone resection, radiation or chemotherapy within past 5 years. Patients with treated basal cell carcinoma or fully cured squamous cell carcinoma are allowed.
2. Any other nasal and sinusoidal diseases or conditions by discretion of the investigator (i.e. nasal polyps, frequent nose bleeding) which may influence the study results
3. Respiratory tract infection or asthma exacerbation in the 4 weeks prior to Visit 1 or during the screening and baseline period.
4. Thoracotomy with pulmonary resection.
5. Previous participation in this study (receipt of randomized treatment) or active participation in a current interventional study.
6. Patients with a clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis at screening, if the abnormality defines a significant disease as defined in exclusion criterion No. 1. Patients will not be randomised if they have increased liver transaminases (AST or ALT greater than two fold the upper limit of normal at screening). Laboratory testing may be repeated once before randomization.
7. Significant alcohol or drug abuse within past 2 years (see exclusion criteria No. 1)
8. Patients with known hypersensitivity to any component of the investigational treatment (see section 4.1.1) or to fluticasone propionate nasal spray or montelukast or salbutamol or components.
9. Patients taking CYP2C8 substrates such as -but not restricted to- amiodarone, amodiaquine, paclitaxel, rosiglitazone, pioglitazone, and repaglinide and CYP2C9 substrates such as -but not restricted to- warfarin, tolbutamide, phenytoin, losartan and acenocoumarol.
10. Patients who have been treated with any of the following medications in the given interval before the respective Visit: Before Visit 2

    * An investigational drug within 1 month or six half lives (whichever is greater)
    * Any immunomodulatory therapy since specific positive skin prick test.
    * A biological based antagonist therapy including Omalizumab, or immune modulator therapy within 6 months
    * A systemic (intravenous, intramuscular or oral) corticosteroid within 3 months
    * The following medications within 4 weeks: topical steroids, change in prescription medications
    * The following medications within 2 weeks: LABA (long acting beta agonist), methylxanthines, leukotriene modifiers, any antihistamines, oral decongestants, any anti-rhinitis therapies (i.e., decongestants, herbals, anticholinergics), and hay-fever medications, tricyclic antidepressants, aspirin and any NSAIDs (non steroidal anti inflammatory drugs) (for occasional pain relief, only paracetamol may be used), oral beta 2 agonists
    * Before Visit 1: Short acting bronchodilator within 6 hours of baseline pulmonary function testing
11. Patients with a risk for prolonged QT interval effects including:

    * A marked baseline prolongation of the QT interval in the electrocardiogram by demonstration of a QTcB interval (Bazett's correction formula) > 450 ms
    * A history of additional risk factors for TdP (Torsades de pointes) e.g., heart failure, hypokalemia, family, history of Long QT Syndrome, etc.
    * The use of concomitant medications known to prolong the QT/QTc interval
12. Pregnant or nursing women
13. Women of childbearing potential not using a highly effective method of birth control.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) as AUC (area under the curve) of values over the entire period from 0-6 hours (h) in the ECC (Environmental Challenge Chamber) | After 2 wks of active treatment compared to 2 wks treatment with placebo

SECONDARY OUTCOMES:
Total Symptom Score (TSSc) as AUC of values for the following periods: 0-2h; 2-4h; 4-6h; 2-6h; 0-6h; 0h-tmax; tmax-6h and hourly | After 2 wks of active treatment compared to 2 wks treatment with placebo
TNSS as AUC of values for the following periods: 0-2h; 2-4h; 4-6h; 2-6; 0h-tmax; tmax-6h and hourly | After 2 wks of active treatment compared to 2 wks treatment with placebo
Total Ocular Symptom Score (TOSS) as AUC of values for the following periods: 0-2h; 2-4h; 4-6h; 2-6h; 0-6h; 0h-tmax; tmax- 6h and hourly | After 2 wks of active treatment compared to 2 wks treatment with placebo
Nasal and ocular sub-scores (single symptoms of TNSS and TOSS) as AUC of values for the following periods: 0-2h; 2-4h; 4-6h; 2-6h; 0-6h; 0h-tmax; tmax-6h and hourly | After 2 wks of active treatment compared to 2 wks treatment with placebo
Flow rate from rhinomanometry as AUC of values obtained at 2, 4 and 6 h | After 2 wks of active treatment compared to 2 wks treatment with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1268.41.49001 Boehringer Ingelheim Investigational Site, Hanover, Germany

REFERENCES:
- [Derived] Krug N, Gupta A, Badorrek P, Koenen R, Mueller M, Pivovarova A, Hilbert J, Wetzel K, Hohlfeld JM, Wood C. Efficacy of the oral chemoattractant receptor homologous molecule on TH2 cells antagonist BI 671800 in patients with seasonal allergic rhinitis. J Allergy Clin Immunol. 2014 Feb;133(2):414-9. doi: 10.1016/j.jaci.2013.10.013. Epub 2013 Dec 9. PMID 24332218